CLINICAL TRIAL: NCT00103142
Title: A Phase II Study of Active Immunotherapy With PANVAC or Autologous, Cultured Dendritic Cells Infected With PANVAC After Complete Resection of Hepatic or Pulmonary Metastases of Colorectal Carcinoma
Brief Title: Vaccine Therapy in Treating Patients With Liver or Lung Metastases From Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Michael Morse, MD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Michael Morse, MD, Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00007616; DUMC-5883-04-6RO (Other: Legacy Duke IRB Number); CDR000041079 (Other: NCI)
Record Dates: First submitted 2005-02-07; First posted 2005-02-08 (Estimated); Results first posted 2014-04-07 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: liver metastases; adenocarcinoma of the colon; recurrent colon cancer; stage IV colon cancer; adenocarcinoma of the rectum; recurrent rectal cancer; stage IV rectal cancer; lung metastases
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PANVAC-V + PANVAC-F + DC (Experimental): Patients undergo leukapheresis to obtain leukocytes for generation of autologous dendritic cells (DC). Patients then receive autologous DC loaded with vaccinia-CEA-MUC-1-TRICOM (PANVAC-V) vaccine subcutaneously (SC) and intradermally (ID) on day 1 and autologous DC loaded with fowlpox-CEA-MUC-1-TRICOM (PANVAC-F) vaccine SC and ID on days 28, 56, and 84.
  Interventions: Biological: falimarev; Biological: inalimarev; Biological: therapeutic autologous dendritic cells
- PANVAC-V + PANVAC-F + GM-CSF (Experimental): Patients receive PANVAC-V SC on day 1 and PANVAC-F SC on days 28, 56, and 84. Patients also receive sargramostim (GM-CSF) SC into the same injection site once daily on days 0-3, 28-31, 56-59, and 84-87.
  Interventions: Biological: falimarev; Biological: inalimarev; Biological: sargramostim

INTERVENTIONS:
Biological: falimarev — Given subcutaneously and intradermally
Biological: inalimarev — Given subcutaneously and intradermally
Biological: sargramostim — Given subcutaneously
  Arms: PANVAC-V + PANVAC-F + GM-CSF
Biological: therapeutic autologous dendritic cells — Given subcutaneously and intradermally
  Arms: PANVAC-V + PANVAC-F + DC

SUMMARY:
RATIONALE: Vaccines made from a gene-modified virus and a person's white blood cells may make the body build an effective immune response to kill tumor cells. Biological therapies, such as Granulocyte-macrophage colony-stimulating factor (GM-CSF), may stimulate the immune system in different ways and stop tumor cells from growing. Combining different types of biological therapies may kill more tumor cells.

PURPOSE: This randomized phase II trial is studying giving vaccine therapy together with dendritic cells to see how well it works compared to giving vaccine therapy together with GM-CSF in treating patients with liver or lung metastases from colorectal cancer removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare 2-year disease-free survival of patients with completely resected hepatic or pulmonary metastases secondary to colorectal cancer treated with adjuvant vaccine therapy comprising vaccinia-Carcinoembryonic antigen (CEA)-mucin 1 (MUC-1)- Triad of costimulatory molecules TRICOM vaccine (PANVAC-V) and fowlpox-CEA-MUC-1-TRICOM vaccine (PANVAC-F) administered with autologous dendritic cells or with sargramostim (GM-CSF).

Secondary

* Compare the rate and magnitude of immune response, as determined by enzyme-linked immunosorbent spot (ELISpot), in patients treated with these regimens.

OUTLINE: This is a randomized study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo leukapheresis to obtain leukocytes for generation of autologous dendritic cells (DC). Patients then receive autologous DC loaded with vaccinia-CEA-MUC-1-TRICOM (PANVAC-V) vaccine subcutaneously (SC) and intradermally (ID) on day 1 and autologous DC loaded with fowlpox-CEA-MUC-1-TRICOM (PANVAC-F) vaccine subcutaneously (SC) and intradermally (ID) on days 28, 56, and 84.
* Arm II: Patients receive PANVAC-V SC on day 1 and PANVAC-F SC on days 28, 56, and 84. Patients also receive sargramostim (GM-CSF) SC into the same injection site once daily on days 0-3, 28-31, 56-59, and 84-87.

After completion of study treatment, patients are followed for 2 years.

PROJECTED ACCRUAL: A total of 72 patients (36 per treatment arm) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed hepatic or pulmonary metastases secondary to adenocarcinoma of the colon and rectum
* Must have undergone complete resection of hepatic or pulmonary metastases with curative intent

  * No evidence of gross residual disease after surgery
  * One or more resected and ablated lesions allowed provided all gross residual tumor was destroyed by ablation
  * Repeated resections of hepatic metastatic disease or resections of extrahepatic metastases prior to resection of the hepatic metastases allowed provided the most recent hepatic metastatic resection included total disease resection and/or ablation
* Must have received at least 2 months of perioperative systemic chemotherapy (including preoperative and/or postoperative chemotherapy) that was completed at least 1 month ago

PATIENT CHARACTERISTICS:

Age

* At least 18

Performance status

* Karnofsky 70-100%

Life expectancy

* At least 6 months

Hematopoietic

* Platelet count ≥ 75,000/mm^3
* Hemoglobin ≥ 8.5 g/dL (transfusion or epoetin alfa allowed)

Hepatic

* Bilirubin ≤ 2.0 mg/dL
* Hepatitis B surface antigen negative
* Hepatitis C antibody negative
* No other serious chronic or acute hepatic disease

Renal

* Creatinine ≤ 1.5 mg/dL OR
* Creatinine clearance > 60 mL/min

Cardiovascular

* No New York Heart Association class III or IV cardiac disease
* No other serious chronic or acute cardiac disease

Pulmonary

* No asthma
* No chronic obstructive pulmonary disease
* No other serious chronic or acute pulmonary disease

Immunologic

* No history of autoimmune disease, including, but not limited to, any of the following:

  * Inflammatory bowel disease
  * Systemic lupus erythematosus
  * Ankylosing spondylitis
  * Scleroderma
  * Multiple sclerosis
* No human immunodeficiency virus (HIV) infection by enzyme-linked immunosorbent assay (ELISA) and western blot
* Not immunocompromised (by disease or therapy)
* No allergy to eggs or any component of the study vaccine
* No history of allergy or untoward reaction to prior vaccinia (smallpox) vaccination
* No allergy or untoward reaction to sargramostim (GM-CSF)
* No active acute or chronic infection, including urinary tract infection within the past 72 hours
* No inflammatory bowel conditions, including, but not limited to, the following:

  * Active infectious enteritis
  * Eosinophilic enteritis
* No acute, chronic, or exfoliative skin disorders, including any of the following:

  * Extensive psoriasis
  * Burns
  * Impetigo
  * Disseminated zoster
  * Varicella zoster
  * Severe acne
  * Other open rashes or wounds

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* Able to avoid close contact or household contact for 3 weeks after each vaccination with the following individuals:

  * Children under 5 years of age
  * Pregnant or nursing women
  * Individuals with prior or concurrent extensive eczema, other eczematoid skin disorders, or other acute or chronic skin conditions
  * Immunosuppressed or immunodeficient individuals
* No medical or psychological condition that would preclude study compliance
* No extensive eczema
* No other serious chronic or acute illness that would preclude study participation
* No other malignancy within the past 5 years except nonmelanoma skin cancer, controlled superficial bladder cancer, or previously treated carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No other concurrent immunotherapy

Chemotherapy

* See Disease Characteristics
* No concurrent chemotherapy

Endocrine therapy

* More than 6 weeks since prior and no concurrent steroid therapy

Radiotherapy

* No concurrent radiotherapy

Surgery

* See Disease Characteristics

Other

* No other concurrent immunosuppressants (e.g., azathioprine or cyclosporine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2005-02; Primary Completion 2009-06 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Morse, MD, Study Chair — Duke Cancer Institute
Locations (6):
- United States (6):
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina

REFERENCES:
- [Derived] Morse MA, Niedzwiecki D, Marshall JL, Garrett C, Chang DZ, Aklilu M, Crocenzi TS, Cole DJ, Dessureault S, Hobeika AC, Osada T, Onaitis M, Clary BM, Hsu D, Devi GR, Bulusu A, Annechiarico RP, Chadaram V, Clay TM, Lyerly HK. A randomized phase II study of immunization with dendritic cells modified with poxvectors encoding CEA and MUC1 compared with the same poxvectors plus GM-CSF for resected metastatic colorectal cancer. Ann Surg. 2013 Dec;258(6):879-86. doi: 10.1097/SLA.0b013e318292919e. PMID 23657083

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 7 site study where patients were recruited from medical clinics and the patient's primary oncologist and study team approached the patient about the study. Patients were recruited for this study from January 2005 and September 2009.
Pre-assignment Details: The study was designed to treat 72 subjects. Total number of enrollment is 74 because enrollment reflects the number of subjects that signed consent and were randomized to the study but did not necessarily receive study drug or complete study drug.
Period: Overall Study
Arm/Group | PANVAC-V + PANVAC-F + DC | PANVAC-V + PANVAC-F + GM-CSF
Started | 36 | 37
Completed | 33 | 36
Not Completed | 3 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Progression of disease | 2 | 1

BASELINE CHARACTERISTICS:
Population: 37 PANVAC-V + PANVAC-F + DC arm patients and 37 PANVAC-V + PANVAC-F + GM-CSF arm. One participant in PANVAC-V + PANVAC-F + DC Arm was consented and contributed baseline data, but was not considered to have started or enrolled in the study patients signed consent.
Groups:
- Experimental PANVAC-V + PANVAC-F + DC: Patients undergo leukapheresis to obtain leukocytes for generation of autologous dendritic cells (DC). Patients then receive autologous DC loaded with vaccinia-Carcinoembryonic antigen (CEA)-Mucin 1 (MUC-1)-TRIad of COstimulatory Molecules (TRICOM) (PANVAC-V) vaccine subcutaneously (SC) and intradermally (ID) on day 1 and autologous DC loaded with fowlpox-CEA-MUC-1-TRICOM (PANVAC-F) vaccine subcutaneous (SC) and intradermally (ID) on days 28, 56, and 84.
- Experimental PANVAC-V + PANVAC-F + GM-CSF: Patients receive PANVAC-V SC on day 1 and PANVAC-F SC on days 28, 56, and 84. Patients also receive sargramostim (Granulocyte-macrophage colony-stimulating factor or GM-CSF) subcutaneous (SC) into the same injection site once daily on days 0-3, 28-31, 56-59, and 84-87.
- Total: Total of all reporting groups
Arm/Group | Experimental PANVAC-V + PANVAC-F + DC | Experimental PANVAC-V + PANVAC-F + GM-CSF | Total
Number analyzed (Participants) | 37 | 37 | 74
Age, Continuous [Median (Full Range); unit: years] | 53.6 [25 to 77] | 52.0 [33 to 74] | 53.5 [25 to 77]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 30 | 58
  >=65 years | 9 | 7 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 18 | 39
  Male | 16 | 19 | 35
Region of Enrollment [Number; unit: participants]
  United States | 37 | 37 | 74
Sites of metastasis [Number; unit: participants]
  Liver | 26 | 31 | 57
  Lung | 11 | 6 | 17
Number of nodules [Number; unit: participants]
  1 nodules | 11 | 17 | 28
  2-4 nodules | 16 | 12 | 28
  >4 nodules | 4 | 5 | 9
  unknown | 6 | 3 | 9
Carcinoembryonic antigen (CEA) [Mean (Full Range); unit: mcg/L] | 2.0 [0.6 to 13.0] | 1.8 [0.5 to 15.0] | 1.9 [0.5 to 15.0]

OUTCOME MEASURES:

1. Primary Outcome: Recurrence-free Survival at 2 Years
Description: Recurrence-free survival for randomized patients receiving dendritic cells (DC) loaded with PANVAC or PANVAC plus Granulocyte-macrophage colony-stimulating factor (GM-CSF) measured from the date of metastasectomy, with relapse defined as documented disease recurrence at any site.
Time Frame: 2 years
Measure: Number; unit: participants
Groups:
- PANVAC-V + PANVAC-F + DC: Patients undergo leukapheresis to obtain leukocytes for generation of autologous dendritic cells (DC). Patients then receive autologous DC loaded with vaccinia-carcinoembryonic antigen (CEA)- mucin 1 (MUC-1)-TRiad of Costimulatory Molecules (TRICOM) (PANVAC-V) vaccine subcutaneously (SC) and intradermally (ID) on day 1 and autologous DC loaded with fowlpox-CEA-MUC-1-TRICOM (PANVAC-F) vaccine subcutaneously (SC) and intradermally (ID) on days 28, 56, and 84.
- PANVAC-V + PANVAC-F + GM-CSF: Patients receive PANVAC-V SC on day 1 and PANVAC-F SC on days 28, 56, and 84. Patients also receive sargramostim (GM-CSF) subcutaneously (SC) into the same injection site once daily on days 0-3, 28-31, 56-59, and 84-87.
Arm/Group | PANVAC-V + PANVAC-F + DC | PANVAC-V + PANVAC-F + GM-CSF
Number analyzed (Participants) | 16 | 20
participants | 13 | 10

2. Secondary Outcome: Positive Immune Response as Measured by (Enzyme-linked Immunosorbent Spot) ELISpot Assay
Description: CEA-Specific Immune Responders by enzyme-linked immunosorbent spot (ELISpot). The ELISPOT assay is considered positive for a subject if the mean number of spots with CEA exceeds the number of spots with control by a magnitude of 10 and the difference between CEA and control is statistically significant at a level of p=0.05 by the t-test.
Time Frame: 13 weeks
Measure: Number; unit: participants
Arm/Group | PANVAC-V + PANVAC-F + DC | PANVAC-V + PANVAC-F + GM-CSF
Number analyzed (Participants) | 35 | 32
participants | 9 | 4

ADVERSE EVENTS:
Description: Adverse Events were only collected/assessed for participants who received at least one dose of intervention
Groups:
- Arm I: Patients undergo leukapheresis to obtain leukocytes for generation of autologous dendritic cells (DC). Patients then receive autologous DC loaded with vaccinia-CEA-MUC-1-TRICOM (PANVAC-V) vaccine subcutaneously (SC) and intradermally (ID) on day 1 and autologous DC loaded with fowlpox-CEA-MUC-1-TRICOM (PANVAC-F) vaccine SC and ID on days 28, 56, and 84.
- Arm II: Patients receive PANVAC-V SC on day 1 and PANVAC-F SC on days 28, 56, and 84. Patients also receive sargramostim (GM-CSF) SC into the same injection site once daily on days 0-3, 28-31, 56-59, and 84-87.
Arm/Group | Arm I | Arm II
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/36
Other Adverse Events (participants affected / at risk) | 35/35 | 35/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=35) | Arm II (N=36)
Hematologic Adverse Events (Blood and lymphatic system disorders) | 8 (8) | 8 (9) — Hematologic Adverse Events
Cardiac (Cardiac disorders) | 1 (1) | 5 (5) — Cardiac
CONSTITUTIONAL SYMPTOMS (General disorders) | 18 (18) | 13 (13) — CONSTITUTIONAL SYMPTOMS
Skin (Skin and subcutaneous tissue disorders) | 30 (30) | 23 (23) — Skin
Endocrine (Endocrine disorders) | 1 (1) | 0 (0) — Endocrine
GI (Gastrointestinal disorders) | 5 (5) | 8 (8) — GI
Infection (Infections and infestations) | 0 (0) | 1 (1) — Infection
Metabolic (Metabolism and nutrition disorders) | 14 (14) | 9 (9)
MUSCULOSKELETAL/SOFT TISSUE (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
NEUROLOGY (Nervous system disorders) | 7 (7) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No